CLINICAL TRIAL: NCT02386371
Title: Feasibility Clinical Trial of Intraoperative Radiotherapy (IORT) and Second Breast-conserving-surgery After Local Recurrence of Breast Carcinoma
Brief Title: Intraoperative Radiotherapy After Local Recurrence in Breast Cancer
Acronym: RE-IORT01
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut du Cancer de Montpellier - Val d'Aurelle (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ICM-URC2014/07
Record Dates: First submitted 2015-03-02; First posted 2015-03-11 (Estimated); Results first posted 2025-02-06 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-02

CONDITIONS: Breast Carcinoma
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- surgery and Intra Operative Radiotherapy (Experimental): Surgery :
  Tumorectomy will be performed according to the current standards, obtaining "clear" margins. The axillary lymph node control will depend on the initial management (clinical and ultrasound) of these N0 patients, chosen by the teams.
  Intra Operative Radiotherapy (IORT):
  After the excision of the tumor, IORT will be delivered. A single dose of 20 Gy by 50 kV photons (Intrabeam™) will be administered in tumor bed. The addition of IORT does not modify the surgical procedure.
  Interventions: Procedure: tumorectomy; Radiation: Intra Operative Radiotherapy

INTERVENTIONS:
Procedure: tumorectomy — Tumorectomy will be performed according to the current standards, obtaining "clear" margins. The axillary lymph node control will depend on the initial management (clinical and ultrasound) of these N0 patients, chosen by the teams.
Radiation: Intra Operative Radiotherapy — After the excision of the tumor, IORT will be delivered. A single dose of 20 Gy by 50 kV photons (Intrabeam™) will be administered in tumor bed. The addition of IORT does not modify the surgical procedure

SUMMARY:
The investigators propose a prospective, multicenter, single arm Phase II design to evaluate the feasibility of repeated breast-conserving surgery combined with re- irradiation using IORT after local recurrence of breast carcinoma.

DETAILED DESCRIPTION:
Currently, the rate of ipsilateral breast tumor recurrence (IBTR) after breast- conserving surgery and radiotherapy remains at 10% at 10 years to 15% at 20 years, respectively. IBTR is an independent predictor of poor survival with a 3 to 4.6 increased risk of cancer-related death.

In a heterogeneous population, local control remains a major therapeutic challenge for these relapses, especially those considered of better prognosis, namely occurring late and of low histological grade. Therapeutic de-escalation is possible for these relapses to avoid a mutilating and often traumatic mastectomy.

However, this second conservative surgery has a high rate of second local relapse (19 to 50% at 5 years) due to the absence of a re-irradiation, rendered impossible by the problem of tolerance of previously irradiated tissues.

Retrospective or prospective studies on partial breast irradiation (PBI) in adjuvant setting report promising results, both in terms of tolerance (saving healthy tissue) and local control (74% to 100% at 5 years). Used techniques include brachytherapy, external beam radiotherapy and intraoperative radiotherapy (IORT).

IORT is now the subject of renewed interest in breast cancer. It has the advantages of high-precision ballistics on the operated area and of preservation of healthy tissue. To date, no prospective data, however, have been published in the indication of ipsilateral breast recurrence.

A prospective, multicenter, single arm Phase II design will evaluate the feasibility of repeated breast-conserving surgery combined with re- irradiation using IORT after local recurrence of breast carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven non-lobular invasive breast recurrence
* Time from whole breast radiation following the initial lumpectomy >5 years
* Unifocal tumor
* Recurrent tumor size ≤ 2 cm
* Adequate breast size for a second breast-conserving surgery with acceptable cosmetic result
* Bilateral breast mammogram within 90 days prior to study entry
* Breast MRI within 90 days prior to study entry
* Histological grade I-II
* Estrogen-receptor-positive tumor (ER+)
* Cerb2-negative tumor
* N0
* M0
* Prior radiotherapy delivered within a standard fractionation schedule
* Performance status (ECOG) 0-1
* Women ≥ 50 years -Absence of any psychological, familial, sociological, or geographical conditions with a potential to hamper compliance with the study and follow- up schedule
* Affiliated to the French Health Insurance regimen
* Written and signed informed consent form.

Exclusion Criteria:

* Multifocal and/or multicenter recurrence
* Lobular carcinoma
* Estrogen-receptor-negative tumor (ER-)
* Cerb2 (her2) overexpressed - breast cancer
* Extensive intraductal component (EIC) on biopsy
* Lymph vessel invasion on biopsy
* N1-3 status: Regional cytological or histologically proven node recurrence
* M1 status: Metastatic disease
* cT4 (Skin or muscle involvement) or Paget's disease of the nipple
* Prior radiotherapy delivered within an accelerated or hypo-fraction schedule
* Prior malignancy other than non-melanoma skin cancer unless the patient has been disease free for at least 5 years
* Patients with a small breast volume, technically unsatisfactory for a second conservative surgery or intraoperative breast irradiation.
* Preoperative chemotherapy or hormone therapy for local relapse
* Connective tissue disease or scleroderma, contraindicating radiotherapy
* Known BRCA1/2 gene mutation (genetic testing is not required)

Min Age: 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2014-03 (Actual); Primary Completion 2020-06-12 (Actual); Study Completion 2023-09-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: LEMANSKI Claire, Study Chair — Institut régional du Cancer - Val d'Aurelle
Locations (8):
- France (8):
  - Institut Bergonié, Bordeaux
  - Chu Brest, Brest
  - Centre George Francois Leclerc, Dijon
  - Centre Léon Bérard, Lyon
  - CHU La TIMONE, Marseille
  - Institut Paoli Calmette, Marseille
  - ICM, Montpellier
  - Institut de Cancérologie de l'Ouest, Nantes

REFERENCES:
- [Background] Fisher B, Anderson S, Bryant J, Margolese RG, Deutsch M, Fisher ER, Jeong JH, Wolmark N. Twenty-year follow-up of a randomized trial comparing total mastectomy, lumpectomy, and lumpectomy plus irradiation for the treatment of invasive breast cancer. N Engl J Med. 2002 Oct 17;347(16):1233-41. doi: 10.1056/NEJMoa022152. PMID 12393820
- [Background] Veronesi U, Cascinelli N, Mariani L, Greco M, Saccozzi R, Luini A, Aguilar M, Marubini E. Twenty-year follow-up of a randomized study comparing breast-conserving surgery with radical mastectomy for early breast cancer. N Engl J Med. 2002 Oct 17;347(16):1227-32. doi: 10.1056/NEJMoa020989. PMID 12393819
- [Background] Brewster AM, Hortobagyi GN, Broglio KR, Kau SW, Santa-Maria CA, Arun B, Buzdar AU, Booser DJ, Valero V, Bondy M, Esteva FJ. Residual risk of breast cancer recurrence 5 years after adjuvant therapy. J Natl Cancer Inst. 2008 Aug 20;100(16):1179-83. doi: 10.1093/jnci/djn233. Epub 2008 Aug 11. PMID 18695137
- [Background] Panet-Raymond V, Truong PT, Alexander C, Lesperance M, McDonald RE, Watson PH. Clinicopathologic factors of the recurrent tumor predict outcome in patients with ipsilateral breast tumor recurrence. Cancer. 2011 May 15;117(10):2035-43. doi: 10.1002/cncr.25767. Epub 2010 Nov 29. PMID 21523714
- [Background] Early Breast Cancer Trialists' Collaborative Group (EBCTCG); Darby S, McGale P, Correa C, Taylor C, Arriagada R, Clarke M, Cutter D, Davies C, Ewertz M, Godwin J, Gray R, Pierce L, Whelan T, Wang Y, Peto R. Effect of radiotherapy after breast-conserving surgery on 10-year recurrence and 15-year breast cancer death: meta-analysis of individual patient data for 10,801 women in 17 randomised trials. Lancet. 2011 Nov 12;378(9804):1707-16. doi: 10.1016/S0140-6736(11)61629-2. Epub 2011 Oct 19. PMID 22019144
- [Background] Kurtz JM, Spitalier JM, Amalric R, Brandone H, Ayme Y, Jacquemier J, Hans D, Bressac C. The prognostic significance of late local recurrence after breast-conserving therapy. Int J Radiat Oncol Biol Phys. 1990 Jan;18(1):87-93. doi: 10.1016/0360-3016(90)90271-k. PMID 2298639
- [Background] Hannoun-Levi JM, Resch A, Gal J, Kauer-Dorner D, Strnad V, Niehoff P, Loessl K, Kovacs G, Van Limbergen E, Polgar C; GEC-ESTRO Breast Cancer Working Group. Accelerated partial breast irradiation with interstitial brachytherapy as second conservative treatment for ipsilateral breast tumour recurrence: multicentric study of the GEC-ESTRO Breast Cancer Working Group. Radiother Oncol. 2013 Aug;108(2):226-31. doi: 10.1016/j.radonc.2013.03.026. Epub 2013 May 3. PMID 23647758
- [Background] Moran MS, Haffty BG. Local-regional breast cancer recurrence: prognostic groups based on patterns of failure. Breast J. 2002 Mar-Apr;8(2):81-7. doi: 10.1046/j.1524-4741.2002.08202.x. PMID 11896752
- [Background] Fourquet A, Campana F, Zafrani B, Mosseri V, Vielh P, Durand JC, Vilcoq JR. Prognostic factors of breast recurrence in the conservative management of early breast cancer: a 25-year follow-up. Int J Radiat Oncol Biol Phys. 1989 Oct;17(4):719-25. doi: 10.1016/0360-3016(89)90057-6. PMID 2777661
- [Background] Fisher B, Anderson S, Fisher ER, Redmond C, Wickerham DL, Wolmark N, Mamounas EP, Deutsch M, Margolese R. Significance of ipsilateral breast tumour recurrence after lumpectomy. Lancet. 1991 Aug 10;338(8763):327-31. doi: 10.1016/0140-6736(91)90475-5. PMID 1677695
- [Background] Veronesi U, Marubini E, Del Vecchio M, Manzari A, Andreola S, Greco M, Luini A, Merson M, Saccozzi R, Rilke F, et al. Local recurrences and distant metastases after conservative breast cancer treatments: partly independent events. J Natl Cancer Inst. 1995 Jan 4;87(1):19-27. doi: 10.1093/jnci/87.1.19. PMID 7666458
- [Background] Tanis E, van de Velde CJ, Bartelink H, van de Vijver MJ, Putter H, van der Hage JA. Locoregional recurrence after breast-conserving therapy remains an independent prognostic factor even after an event free interval of 10 years in early stage breast cancer. Eur J Cancer. 2012 Aug;48(12):1751-6. doi: 10.1016/j.ejca.2012.02.051. Epub 2012 Mar 23. PMID 22446021
- [Background] Schmoor C, Sauerbrei W, Bastert G, Schumacher M. Role of isolated locoregional recurrence of breast cancer: results of four prospective studies. J Clin Oncol. 2000 Apr;18(8):1696-708. doi: 10.1200/JCO.2000.18.8.1696. PMID 10764430
- [Background] Anderson SJ, Wapnir I, Dignam JJ, Fisher B, Mamounas EP, Jeong JH, Geyer CE Jr, Wickerham DL, Costantino JP, Wolmark N. Prognosis after ipsilateral breast tumor recurrence and locoregional recurrences in patients treated by breast-conserving therapy in five National Surgical Adjuvant Breast and Bowel Project protocols of node-negative breast cancer. J Clin Oncol. 2009 May 20;27(15):2466-73. doi: 10.1200/JCO.2008.19.8424. Epub 2009 Apr 6. PMID 19349544
- [Background] van der Sangen MJ, van de Poll-Franse LV, Roumen RM, Rutten HJ, Coebergh JW, Vreugdenhil G, Voogd AC. The prognosis of patients with local recurrence more than five years after breast conservation therapy for invasive breast carcinoma. Eur J Surg Oncol. 2006 Feb;32(1):34-8. doi: 10.1016/j.ejso.2005.10.005. Epub 2005 Nov 21. PMID 16305821
- [Background] Galper S, Blood E, Gelman R, Abner A, Recht A, Kohli A, Wong JS, Smith D, Bellon J, Connolly J, Schnitt S, Winer E, Silver B, Harris JR. Prognosis after local recurrence after conservative surgery and radiation for early-stage breast cancer. Int J Radiat Oncol Biol Phys. 2005 Feb 1;61(2):348-57. doi: 10.1016/j.ijrobp.2004.06.011. PMID 15667952
- [Background] Le MG, Arriagada R, Spielmann M, Guinebretiere JM, Rochard F. Prognostic factors for death after an isolated local recurrence in patients with early-stage breast carcinoma. Cancer. 2002 Jun 1;94(11):2813-20. doi: 10.1002/cncr.10572. PMID 12115367
- [Background] Courdi A, Doyen J, Gal J, Chamorey E. Local recurrence after breast cancer affects specific survival differently according to patient age. Oncology. 2010;79(5-6):349-54. doi: 10.1159/000323483. Epub 2011 Mar 23. PMID 21430403
- [Background] Livi L, Meattini I, Marrazzo L, Simontacchi G, Pallotta S, Saieva C, Paiar F, Scotti V, De Luca Cardillo C, Bastiani P, Orzalesi L, Casella D, Sanchez L, Nori J, Fambrini M, Bianchi S. Accelerated partial breast irradiation using intensity-modulated radiotherapy versus whole breast irradiation: 5-year survival analysis of a phase 3 randomised controlled trial. Eur J Cancer. 2015 Mar;51(4):451-463. doi: 10.1016/j.ejca.2014.12.013. Epub 2015 Jan 17. PMID 25605582
- [Background] Sabatier R, Finetti P, Cervera N, Tallet A, Benchalal M, Houvenaeghel G, Jacquemier J, Birnbaum D, Bertucci F. Gene expression profiling and its utility in prediction of local relapse after breast-conserving therapy in early breast cancer. Cancer Genomics Proteomics. 2011 Jul-Aug;8(4):199-209. PMID 21737613
- [Background] Kurtz JM, Jacquemier J, Amalric R, Brandone H, Ayme Y, Hans D, Bressac C, Spitalier JM. Is breast conservation after local recurrence feasible? Eur J Cancer. 1991;27(3):240-4. doi: 10.1016/0277-5379(91)90505-8. PMID 1827303
- [Background] Salvadori B, Marubini E, Miceli R, Conti AR, Cusumano F, Andreola S, Zucali R, Veronesi U. Reoperation for locally recurrent breast cancer in patients previously treated with conservative surgery. Br J Surg. 1999 Jan;86(1):84-7. doi: 10.1046/j.1365-2168.1999.00961.x. PMID 10027366
- [Background] Alpert TE, Kuerer HM, Arthur DW, Lannin DR, Haffty BG. Ipsilateral breast tumor recurrence after breast conservation therapy: outcomes of salvage mastectomy vs. salvage breast-conserving surgery and prognostic factors for salvage breast preservation. Int J Radiat Oncol Biol Phys. 2005 Nov 1;63(3):845-51. doi: 10.1016/j.ijrobp.2005.02.035. PMID 16199315
- [Background] Gentilini O, Botteri E, Veronesi P, Sangalli C, Del Castillo A, Ballardini B, Galimberti V, Rietjens M, Colleoni M, Luini A, Veronesi U. Repeating conservative surgery after ipsilateral breast tumor reappearance: criteria for selecting the best candidates. Ann Surg Oncol. 2012 Nov;19(12):3771-6. doi: 10.1245/s10434-012-2404-5. Epub 2012 May 23. PMID 22618719
- [Background] Deutsch M. Repeat high-dose external beam irradiation for in-breast tumor recurrence after previous lumpectomy and whole breast irradiation. Int J Radiat Oncol Biol Phys. 2002 Jul 1;53(3):687-91. doi: 10.1016/s0360-3016(02)02785-2. PMID 12062613
- [Background] Hannoun-Levi JM, Ihrai T, Courdi A. Local treatment options for ipsilateral breast tumour recurrence. Cancer Treat Rev. 2013 Nov;39(7):737-41. doi: 10.1016/j.ctrv.2013.02.003. Epub 2013 Mar 5. PMID 23465859
- [Background] Chadha M, Feldman S, Boolbol S, Wang L, Harrison LB. The feasibility of a second lumpectomy and breast brachytherapy for localized cancer in a breast previously treated with lumpectomy and radiation therapy for breast cancer. Brachytherapy. 2008 Jan-Mar;7(1):22-8. doi: 10.1016/j.brachy.2007.10.006. PMID 18299110
- [Background] Trombetta M, Julian TB, Werts ED, Colonias A, Betler J, Kotinsley K, Kim Y, Parda D. Comparison of conservative management techniques in the re-treatment of ipsilateral breast tumor recurrence. Brachytherapy. 2011 Jan-Feb;10(1):74-80. doi: 10.1016/j.brachy.2010.01.005. Epub 2010 Aug 4. PMID 20685174
- [Background] Wapnir IL, Aebi S, Gelber S, Anderson SJ, Lang I, Robidoux A, Mamounas EP, Wolmark N. Progress on BIG 1-02/IBCSG 27-02/NSABP B-37, a prospective randomized trial evaluating chemotherapy after local therapy for isolated locoregional recurrences of breast cancer. Ann Surg Oncol. 2008 Nov;15(11):3227-31. doi: 10.1245/s10434-008-0129-2. Epub 2008 Sep 11. PMID 18784962
- [Background] Aebi S, Gelber S, Anderson SJ, Lang I, Robidoux A, Martin M, Nortier JW, Paterson AH, Rimawi MF, Canada JM, Thurlimann B, Murray E, Mamounas EP, Geyer CE Jr, Price KN, Coates AS, Gelber RD, Rastogi P, Wolmark N, Wapnir IL; CALOR investigators. Chemotherapy for isolated locoregional recurrence of breast cancer (CALOR): a randomised trial. Lancet Oncol. 2014 Feb;15(2):156-63. doi: 10.1016/S1470-2045(13)70589-8. Epub 2014 Jan 16. PMID 24439313
- [Background] Borner M, Bacchi M, Goldhirsch A, Greiner R, Harder F, Castiglione M, Jungi WF, Thurlimann B, Cavalli F, Obrecht JP, et al. First isolated locoregional recurrence following mastectomy for breast cancer: results of a phase III multicenter study comparing systemic treatment with observation after excision and radiation. Swiss Group for Clinical Cancer Research. J Clin Oncol. 1994 Oct;12(10):2071-7. doi: 10.1200/JCO.1994.12.10.2071. PMID 7931476
- [Background] Waeber M, Castiglione-Gertsch M, Dietrich D, Thurlimann B, Goldhirsch A, Brunner KW, Borner MM; Swiss Group for Clinical Cancer Research (SAKK). Adjuvant therapy after excision and radiation of isolated postmastectomy locoregional breast cancer recurrence: definitive results of a phase III randomized trial (SAKK 23/82) comparing tamoxifen with observation. Ann Oncol. 2003 Aug;14(8):1215-21. doi: 10.1093/annonc/mdg347. PMID 12881382
- [Background] Doyle T, Schultz DJ, Peters C, Harris E, Solin LJ. Long-term results of local recurrence after breast conservation treatment for invasive breast cancer. Int J Radiat Oncol Biol Phys. 2001 Sep 1;51(1):74-80. doi: 10.1016/s0360-3016(01)01625-x. PMID 11516854
- [Background] Abner AL, Recht A, Eberlein T, Come S, Shulman L, Hayes D, Connolly JL, Schnitt SJ, Silver B, Harris JR. Prognosis following salvage mastectomy for recurrence in the breast after conservative surgery and radiation therapy for early-stage breast cancer. J Clin Oncol. 1993 Jan;11(1):44-8. doi: 10.1200/JCO.1993.11.1.44. PMID 8418240
- [Background] Voogd AC, van Tienhoven G, Peterse HL, Crommelin MA, Rutgers EJ, van de Velde CJ, van Geel BN, Slot A, Rodrigus PT, Jobsen JJ, von Meyenfeldt MF, Coebergh JW. Local recurrence after breast conservation therapy for early stage breast carcinoma: detection, treatment, and outcome in 266 patients. Dutch Study Group on Local Recurrence after Breast Conservation (BORST). Cancer. 1999 Jan 15;85(2):437-46. doi: 10.1002/(sici)1097-0142(19990115)85:23.0.co;2-1. PMID 10023713
- [Background] Moran MS, Schnitt SJ, Giuliano AE, Harris JR, Khan SA, Horton J, Klimberg S, Chavez-MacGregor M, Freedman G, Houssami N, Johnson PL, Morrow M; Society of Surgical Oncology; American Society for Radiation Oncology. Society of Surgical Oncology-American Society for Radiation Oncology consensus guideline on margins for breast-conserving surgery with whole-breast irradiation in stages I and II invasive breast cancer. J Clin Oncol. 2014 May 10;32(14):1507-15. doi: 10.1200/JCO.2013.53.3935. Epub 2014 Feb 10. PMID 24516019
- [Background] Dalberg K, Mattsson A, Sandelin K, Rutqvist LE. Outcome of treatment for ipsilateral breast tumor recurrence in early-stage breast cancer. Breast Cancer Res Treat. 1998 May;49(1):69-78. doi: 10.1023/a:1005934513072. PMID 9694613
- [Background] Ishitobi M, Komoike Y, Nakahara S, Motomura K, Koyama H, Inaji H. Repeat lumpectomy for ipsilateral breast tumor recurrence after breast-conserving treatment. Oncology. 2011;81(5-6):381-6. doi: 10.1159/000335265. Epub 2012 Jan 20. PMID 22269927
- [Background] Chen SL, Martinez SR. The survival impact of the choice of surgical procedure after ipsilateral breast cancer recurrence. Am J Surg. 2008 Oct;196(4):495-9. doi: 10.1016/j.amjsurg.2008.06.018. PMID 18809050
- [Background] Holland R, Veling SH, Mravunac M, Hendriks JH. Histologic multifocality of Tis, T1-2 breast carcinomas. Implications for clinical trials of breast-conserving surgery. Cancer. 1985 Sep 1;56(5):979-90. doi: 10.1002/1097-0142(19850901)56:53.0.co;2-n. PMID 2990668
- [Background] Smith TE, Lee D, Turner BC, Carter D, Haffty BG. True recurrence vs. new primary ipsilateral breast tumor relapse: an analysis of clinical and pathologic differences and their implications in natural history, prognoses, and therapeutic management. Int J Radiat Oncol Biol Phys. 2000 Dec 1;48(5):1281-9. doi: 10.1016/s0360-3016(00)01378-x. PMID 11121624
- [Background] Fredriksson I, Liljegren G, Arnesson LG, Emdin SO, Palm-Sjovall M, Fornander T, Holmqvist M, Holmberg L, Frisell J. Local recurrence in the breast after conservative surgery--a study of prognosis and prognostic factors in 391 women. Eur J Cancer. 2002 Sep;38(14):1860-70. doi: 10.1016/s0959-8049(02)00219-8. PMID 12204668
- [Background] Vaidya JS, Joseph DJ, Tobias JS, Bulsara M, Wenz F, Saunders C, Alvarado M, Flyger HL, Massarut S, Eiermann W, Keshtgar M, Dewar J, Kraus-Tiefenbacher U, Sutterlin M, Esserman L, Holtveg HM, Roncadin M, Pigorsch S, Metaxas M, Falzon M, Matthews A, Corica T, Williams NR, Baum M. Targeted intraoperative radiotherapy versus whole breast radiotherapy for breast cancer (TARGIT-A trial): an international, prospective, randomised, non-inferiority phase 3 trial. Lancet. 2010 Jul 10;376(9735):91-102. doi: 10.1016/S0140-6736(10)60837-9. PMID 20570343
- [Background] Smith BD, Arthur DW, Buchholz TA, Haffty BG, Hahn CA, Hardenbergh PH, Julian TB, Marks LB, Todor DA, Vicini FA, Whelan TJ, White J, Wo JY, Harris JR. Accelerated partial breast irradiation consensus statement from the American Society for Radiation Oncology (ASTRO). J Am Coll Surg. 2009 Aug;209(2):269-77. doi: 10.1016/j.jamcollsurg.2009.02.066. Epub 2009 Apr 24. No abstract available. PMID 19632605
- [Background] Polgar C, Van Limbergen E, Potter R, Kovacs G, Polo A, Lyczek J, Hildebrandt G, Niehoff P, Guinot JL, Guedea F, Johansson B, Ott OJ, Major T, Strnad V; GEC-ESTRO breast cancer working group. Patient selection for accelerated partial-breast irradiation (APBI) after breast-conserving surgery: recommendations of the Groupe Europeen de Curietherapie-European Society for Therapeutic Radiology and Oncology (GEC-ESTRO) breast cancer working group based on clinical evidence (2009). Radiother Oncol. 2010 Mar;94(3):264-73. doi: 10.1016/j.radonc.2010.01.014. Epub 2010 Feb 22. PMID 20181402
- [Background] Hannoun-Levi JM, Houvenaeghel G, Ellis S, Teissier E, Alzieu C, Lallement M, Cowen D. Partial breast irradiation as second conservative treatment for local breast cancer recurrence. Int J Radiat Oncol Biol Phys. 2004 Dec 1;60(5):1385-92. doi: 10.1016/j.ijrobp.2004.05.035. PMID 15590169
- [Background] Resch A, Fellner C, Mock U, Handl-Zeller L, Biber E, Seitz W, Potter R. Locally recurrent breast cancer: pulse dose rate brachytherapy for repeat irradiation following lumpectomy-- a second chance to preserve the breast. Radiology. 2002 Dec;225(3):713-8. doi: 10.1148/radiol.2253011913. PMID 12461250
- [Background] Kraus-Tiefenbacher U, Bauer L, Scheda A, Schoeber C, Schaefer J, Steil V, Wenz F. Intraoperative radiotherapy (IORT) is an option for patients with localized breast recurrences after previous external-beam radiotherapy. BMC Cancer. 2007 Sep 14;7:178. doi: 10.1186/1471-2407-7-178. PMID 17854511
- [Background] Kauer-Dorner D, Potter R, Resch A, Handl-Zeller L, Kirchheiner K, Meyer-Schell K, Dorr W. Partial breast irradiation for locally recurrent breast cancer within a second breast conserving treatment: alternative to mastectomy? Results from a prospective trial. Radiother Oncol. 2012 Jan;102(1):96-101. doi: 10.1016/j.radonc.2011.07.020. Epub 2011 Sep 8. PMID 21907439
- [Background] Guix B, Lejarcegui JA, Tello JI, Zanon G, Henriquez I, Finestres F, Martinez A, Fernandez-Ibiza J, Quinzanos L, Palombo P, Encinas X, Guix I. Exeresis and brachytherapy as salvage treatment for local recurrence after conservative treatment for breast cancer: results of a ten-year pilot study. Int J Radiat Oncol Biol Phys. 2010 Nov 1;78(3):804-10. doi: 10.1016/j.ijrobp.2009.08.009. Epub 2010 Jan 26. PMID 20106605
- [Background] Nairz O, Deutschmann H, Kopp M, Wurstbauer K, Kametriser G, Fastner G, Merz F, Reitsamer R, Menzel C, Sedlmayer F. A dosimetric comparison of IORT techniques in limited-stage breast cancer. Strahlenther Onkol. 2006 Jun;182(6):342-8. doi: 10.1007/s00066-006-1580-2. PMID 16703290
- [Background] Herskind C, Griebel J, Kraus-Tiefenbacher U, Wenz F. Sphere of equivalence--a novel target volume concept for intraoperative radiotherapy using low-energy X rays. Int J Radiat Oncol Biol Phys. 2008 Dec 1;72(5):1575-81. doi: 10.1016/j.ijrobp.2008.08.009. PMID 19028280
- [Background] Liu Q, Schneider F, Ma L, Wenz F, Herskind C. Relative Biologic Effectiveness (RBE) of 50 kV X-rays measured in a phantom for intraoperative tumor-bed irradiation. Int J Radiat Oncol Biol Phys. 2013 Mar 15;85(4):1127-33. doi: 10.1016/j.ijrobp.2012.08.005. Epub 2012 Sep 14. PMID 22981707
- [Background] Reitsamer R, Fastner G, Kopp M, Menzel C, Sedlmayer F. Intraoperative radiotherapy for early breast cancer. Lancet. 2010 Oct 2;376(9747):1141; author reply 1143-4. doi: 10.1016/S0140-6736(10)61529-2. No abstract available. PMID 20888980
- [Background] Smith BD, Buchholz TA, Kuerer HM. Intraoperative radiotherapy for early breast cancer. Lancet. 2010 Oct 2;376(9747):1141; author reply 1143-4. doi: 10.1016/S0140-6736(10)61530-9. No abstract available. PMID 20888981
- [Background] Reitsamer R, Sedlmayer F, Kopp M, Kametriser G, Menzel C, Deutschmann H, Nairz O, Hitzl W, Peintinger F. The Salzburg concept of intraoperative radiotherapy for breast cancer: results and considerations. Int J Cancer. 2006 Jun 1;118(11):2882-7. doi: 10.1002/ijc.21727. PMID 16381011
- [Background] Dubois JB, Hay M, Gely S, Saint-Aubert B, Rouanet P, Pujol H. IORT in breast carcinomas. Front Radiat Ther Oncol. 1997;31:131-7. doi: 10.1159/000061160. No abstract available. PMID 9263806
- [Background] Fastner G, Sedlmayer F, Merz F, Deutschmann H, Reitsamer R, Menzel C, Stierle C, Farmini A, Fischer T, Ciabattoni A, Mirri A, Hager E, Reinartz G, Lemanski C, Orecchia R, Valentini V. IORT with electrons as boost strategy during breast conserving therapy in limited stage breast cancer: long term results of an ISIORT pooled analysis. Radiother Oncol. 2013 Aug;108(2):279-86. doi: 10.1016/j.radonc.2013.05.031. Epub 2013 Jul 2. PMID 23830467
- [Background] Lemanski C, Azria D, Thezenas S, Gutowski M, Saint-Aubert B, Rouanet P, Fenoglietto P, Ailleres N, Dubois JB. Intraoperative radiotherapy given as a boost for early breast cancer: long-term clinical and cosmetic results. Int J Radiat Oncol Biol Phys. 2006 Apr 1;64(5):1410-5. doi: 10.1016/j.ijrobp.2005.10.025. Epub 2006 Jan 25. PMID 16442241
- [Background] Lemanski C, Azria D, Gourgon-Bourgade S, Gutowski M, Rouanet P, Saint-Aubert B, Ailleres N, Fenoglietto P, Dubois JB. Intraoperative radiotherapy in early-stage breast cancer: results of the montpellier phase II trial. Int J Radiat Oncol Biol Phys. 2010 Mar 1;76(3):698-703. doi: 10.1016/j.ijrobp.2009.02.039. Epub 2009 May 23. PMID 19467579
- [Background] Welzel G, Boch A, Sperk E, Hofmann F, Kraus-Tiefenbacher U, Gerhardt A, Suetterlin M, Wenz F. Radiation-related quality of life parameters after targeted intraoperative radiotherapy versus whole breast radiotherapy in patients with breast cancer: results from the randomized phase III trial TARGIT-A. Radiat Oncol. 2013 Jan 7;8:9. doi: 10.1186/1748-717X-8-9. PMID 23294485
- [Background] Sperk E, Welzel G, Keller A, Kraus-Tiefenbacher U, Gerhardt A, Sutterlin M, Wenz F. Late radiation toxicity after intraoperative radiotherapy (IORT) for breast cancer: results from the randomized phase III trial TARGIT A. Breast Cancer Res Treat. 2012 Aug;135(1):253-60. doi: 10.1007/s10549-012-2168-4. Epub 2012 Jul 29. PMID 22842984
- [Background] Grobmyer SR, Lightsey JL, Bryant CM, Shaw C, Yeung A, Bhandare N, Hitchingham B, Copeland EM 3rd. Low-kilovoltage, single-dose intraoperative radiation therapy for breast cancer: results and impact on a multidisciplinary breast cancer program. J Am Coll Surg. 2013 Apr;216(4):617-23; discussion 623-4. doi: 10.1016/j.jamcollsurg.2012.12.038. Epub 2013 Feb 14. PMID 23415885
- [Background] Keshtgar MR, Williams NR, Bulsara M, Saunders C, Flyger H, Cardoso JS, Corica T, Bentzon N, Michalopoulos NV, Joseph DJ. Objective assessment of cosmetic outcome after targeted intraoperative radiotherapy in breast cancer: results from a randomised controlled trial. Breast Cancer Res Treat. 2013 Aug;140(3):519-25. doi: 10.1007/s10549-013-2641-8. Epub 2013 Jul 23. PMID 23877341
- [Background] Dubois JB, Gu SD, Hay MH, Gely S, Delard R, Joyeux H, Solassol C, Pujol H. Intra-operative radiation therapy (IORT) with 100 kV X photons. Experience on 170 patients. Pathol Biol (Paris). 1992 Nov;39(9):884-5. No abstract available. PMID 1538921
- [Background] Lemanski C, Azria D, Gourgou-Bourgade S, Ailleres N, Pastant A, Rouanet P, Fenoglietto P, Dubois JB, Gutowski M. Electrons for intraoperative radiotherapy in selected breast-cancer patients: late results of the Montpellier phase II trial. Radiat Oncol. 2013 Aug 1;8:191. doi: 10.1186/1748-717X-8-191. PMID 23902825
- [Background] Neumaier C, Elena S, Grit W, Yasser AM, Uta KT, Anke K, Axel G, Marc S, Frederik W. TARGIT-E(lderly)--prospective phase II study of intraoperative radiotherapy (IORT) in elderly patients with small breast cancer. BMC Cancer. 2012 May 8;12:171. doi: 10.1186/1471-2407-12-171. PMID 22569123
- [Background] Azria D, Belkacemi Y, Romieu G, Gourgou S, Gutowski M, Zaman K, Moscardo CL, Lemanski C, Coelho M, Rosenstein B, Fenoglietto P, Crompton NE, Ozsahin M. Concurrent or sequential adjuvant letrozole and radiotherapy after conservative surgery for early-stage breast cancer (CO-HO-RT): a phase 2 randomised trial. Lancet Oncol. 2010 Mar;11(3):258-65. doi: 10.1016/S1470-2045(10)70013-9. Epub 2010 Feb 6. PMID 20138810
- [Background] Ozsahin M, Crompton NE, Gourgou S, Kramar A, Li L, Shi Y, Sozzi WJ, Zouhair A, Mirimanoff RO, Azria D. CD4 and CD8 T-lymphocyte apoptosis can predict radiation-induced late toxicity: a prospective study in 399 patients. Clin Cancer Res. 2005 Oct 15;11(20):7426-33. doi: 10.1158/1078-0432.CCR-04-2634. PMID 16243816
- [Background] Rothkamm K, Beinke C, Romm H, Badie C, Balagurunathan Y, Barnard S, Bernard N, Boulay-Greene H, Brengues M, De Amicis A, De Sanctis S, Greither R, Herodin F, Jones A, Kabacik S, Knie T, Kulka U, Lista F, Martigne P, Missel A, Moquet J, Oestreicher U, Peinnequin A, Poyot T, Roessler U, Scherthan H, Terbrueggen B, Thierens H, Valente M, Vral A, Zenhausern F, Meineke V, Braselmann H, Abend M. Comparison of established and emerging biodosimetry assays. Radiat Res. 2013 Aug;180(2):111-9. doi: 10.1667/RR3231.1. Epub 2013 Jul 17. PMID 23862692
- [Background] Templin T, Paul S, Amundson SA, Young EF, Barker CA, Wolden SL, Smilenov LB. Radiation-induced micro-RNA expression changes in peripheral blood cells of radiotherapy patients. Int J Radiat Oncol Biol Phys. 2011 Jun 1;80(2):549-57. doi: 10.1016/j.ijrobp.2010.12.061. Epub 2011 Mar 21. PMID 21420249
- [Background] Park SH, Kim MJ, Park BW, Moon HJ, Kwak JY, Kim EK. Impact of preoperative ultrasonography and fine-needle aspiration of axillary lymph nodes on surgical management of primary breast cancer. Ann Surg Oncol. 2011 Mar;18(3):738-44. doi: 10.1245/s10434-010-1347-y. Epub 2010 Oct 2. PMID 20890729
- [Background] MacNeill M, Arnott I, Thomas J. Fine needle aspiration cytology is a valuable adjunct to axillary ultrasound in the preoperative staging of breast cancer. J Clin Pathol. 2011 Jan;64(1):42-6. doi: 10.1136/jcp.2010.083063. Epub 2010 Nov 19. PMID 21097541

RESULTS

PARTICIPANT FLOW:
Groups:
- Surgery and Intra Operative Radiotherapy: Surgery :
  Tumorectomy will be performed according to the current standards, obtaining "clear" margins. The axillary lymph node control will depend on the initial management (clinical and ultrasound) of these N0 patients, chosen by the teams.
  Intra Operative Radiotherapy (IORT):
  After the excision of the tumor, IORT will be delivered. A single dose of 20 Gy by 50 kV photons (Intrabeam™) will be administered in tumor bed. The addition of IORT does not modify the surgical procedure.
  tumorectomy: Tumorectomy will be performed according to the current standards, obtaining "clear" margins. The axillary lymph node control will depend on the initial management (clinical and ultrasound) of these N0 patients, chosen by the teams.
  Intra Operative Radiotherapy: After the excision of the tumor, IORT will be delivered. A single dose of 20 Gy by 50 kV photons (Intrabeam™) will be administered in tumor bed. The addition of IORT does not modify the surgical procedure
Period: Overall Study
Arm/Group | Surgery and Intra Operative Radiotherapy
Started | 66
Completed | 53
Not Completed | 13

BASELINE CHARACTERISTICS:
Arm/Group | Surgery and Intra Operative Radiotherapy
Number analyzed (Participants) | 53
Age, Continuous [Median (Full Range); unit: years] | 68 [50 to 93]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 53
  Male | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: The Tolerance of RIOP (Intra Operative Radiotherapy) in Patients With Delayed Local Recurrences, After a Second Conservative Treatment of Breast Cancer
Description: Fibrosis rate of RIOP grade 2 at 12 months of IORT (Intra Operative Radiotherapy) according to NCI CTCAE v4.0 classification grade 0 is the better outcomes Grade >= 2 is the worse outcomes
Time Frame: Up to 12 months post radiation
Measure: Number; unit: participants
Arm/Group | Surgery and Intra Operative Radiotherapy
Number analyzed (Participants) | 53
participants
  number of patients without fibrosis | 34
  number of patients with fibrosis | 19

2. Secondary Outcome: Rate of Early and Late Toxicities
Description: Rate of Early toxicities (Hematoma, Lymphorrhea, Breast infection) Late toxicities (telangiectasia, breast pain, skin hyperpigmentation, skin ulceration, skin atrophy) grade 0 is the better outcomes
Time Frame: from the baseline to 5 years after treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Surgery and Intra Operative Radiotherapy
Number analyzed (Participants) | 59
Participants
  global toxicities: grade 0 | 4
  global toxicities: grade 1 | 18
  global toxicities: grade 2 | 27
  global toxicities: grade 3 | 10
  global toxicities: Missing data | 0
  Early toxicities: grade 0 | 12
  Early toxicities: grade 1 | 24
  Early toxicities: grade 2 | 17
  Early toxicities: grade 3 | 4
  Early toxicities: Missing data | 2
  Late toxicities: grade 0 | 5
  Late toxicities: grade 1 | 18
  Late toxicities: grade 2 | 24
  Late toxicities: grade 3 | 8
  Late toxicities: Missing data | 4

3. Secondary Outcome: Local Relapse-free Survival
Description: Number of patient with or without the apparition of local relapse
Time Frame: from the baseline to 5 years after treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Surgery and Intra Operative Radiotherapy
Number analyzed (Participants) | 53
Participants
  patient with a local relapse | 2
  patients without local relapse | 51

4. Secondary Outcome: Metastasis Relapse-free Survival
Description: number of patient with and without the apparition of metastatic relapse.
Time Frame: from the baseline to 5 years after treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Surgery and Intra Operative Radiotherapy
Number analyzed (Participants) | 53
Participants
  patient with a metastatic relapse | 1
  patient without a metastatic relapse | 52

5. Secondary Outcome: Disease-free Survival.
Description: Number of patient with and without a relapse
Time Frame: from the baseline to 5 years after treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Surgery and Intra Operative Radiotherapy
Number analyzed (Participants) | 53
Participants
  patients with relapse | 9
  patients without relapse | 44

6. Secondary Outcome: Overall Survival
Description: number de patient dead
Time Frame: from the baseline to 5 years after treatment
Population: only 53 patients analysable for this objective
Measure: Number; unit: participants
Arm/Group | Surgery and Intra Operative Radiotherapy
Number analyzed (Participants) | 53
participants | 6

7. Secondary Outcome: Free Interval Without Mastectomy.
Description: Number of patient with a mastectomy during the study and follow up
Time Frame: from the baseline to 5 years after treatment
Population: number of patient with mastectomy
Measure: Number; unit: participants
Arm/Group | Surgery and Intra Operative Radiotherapy
Number analyzed (Participants) | 53
participants | 3

ADVERSE EVENTS:
Time Frame: adverse event were collected from baseline to 5 years after the surgery
Arm/Group | Surgery and Intra Operative Radiotherapy
All-Cause Mortality (participants affected / at risk) | 6/59
Serious Adverse Events (participants affected / at risk) | 3/59
Other Adverse Events (participants affected / at risk) | 59/59
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Surgery and Intra Operative Radiotherapy (N=59)
lumbosacral radiculopathy (Musculoskeletal and connective tissue disorders) | 1 (1)
postoperative wound infection (Infections and infestations) | 1 (1)
mastitis (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Surgery and Intra Operative Radiotherapy (N=59)
hearing and inner ear disorder (Ear and labyrinth disorders) | 1 (1)
visual system disorder (Eye disorders) | 2 (2)
gastrointestinal disorders (Gastrointestinal disorders) | 4 (4)
general disorders and reaction at the site of administration (General disorders) | 16 (16)
Infections and infestations (Infections and infestations) | 3 (3)
medical exams (Investigations) | 3 (3)
metabolism and nutrition disorders (Metabolism and nutrition disorders) | 2 (2)
musculoskeletal and connective tissue disorders (Musculoskeletal and connective tissue disorders) | 49 (49)
nervous system disorder (Nervous system disorders) | 2 (2)
psychiatric disorders (Psychiatric disorders) | 4 (4)
renal and urinary disorders (Renal and urinary disorders) | 1 (1)
reproductive system and breast disorders (Reproductive system and breast disorders) | 29 (29)
respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 1 (1)
skin and subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 37 (37)
surgical ann medical procedures (Surgical and medical procedures) | 1 (1)
vascular disorders (Vascular disorders) | 25 (25)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol (2017-06-26): https://cdn.clinicaltrials.gov/large-docs/71/NCT02386371/Prot_000.pdf